CLINICAL TRIAL: NCT06820060
Title: An Observational, Prospective and Retrospective Clinical Study to Evaluate the Performance of QIAstat-Dx® Meningitis/Encephalitis (ME) Panel Plus During Normal Conditions of Use
Brief Title: Clinical Performance of QIAstat-Dx® Meningitis/Encephalitis (ME) Panel Plus
Status: Active, not recruiting | Type: Observational
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: DHF-18-0489-1-CSP-003
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-04

CONDITIONS: Meningitis; Encephalitis Infection
Keywords: Meningitis infection; QIAstat-Dx; Clinical Performance Study; Encephalitis infection
MeSH Terms: conditions — Meningitis; Infectious Encephalitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh Cerebrospinal specimens Selected archived frozen specimens will be tested retrospectively if required.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Performance evaluation of QIAstat-Dx® ME Panel Plus using the QIAstat-Dx® Analyzer to demonstrate that the QIAstat-Dx® ME Panel Plus achieves its intended performance during normal conditions of use by the intended user in the intended environment

DETAILED DESCRIPTION:
The objective of the study is to demonstrate that the QIAstat-Dx® ME Panel Plus achieves its intended performance during normal conditions of use by the intended user in the intended environment.

The primary objective is to evaluate the performance of QIAstat-Dx® ME Panel Plus in comparison with the results obtained from the reference method.

The secondary objective of the study is to evaluate the safety of QIAstat-Dx® ME Panel Plus with respect to users/operators.

The primary study endpoint will be the results for each analyte obtained from testing prospective and retrospective specimens with QIAstat-Dx® ME Panel Plus and Reference Method. Positive Percent Agreement (PPA) and Negative Percent Agreement (NPA) will be determined

ELIGIBILITY:
Inclusion Criteria:

* Specimen must be Cerebrospinal fluid, obtained via lumbar puncture only.
* Specimen must be a de-identified residual leftover specimen.
* Specimen must meet the laboratory testing criteria for individuals with signs and/or symptoms of meningitis and/or encephalitis.
* Specimens must have a minimum 450 µL of residual volume.
* Specimen must be unique (only one sample enrolled per patient).
* Prior to QIAstat-Dx testing, residual CSF specimen must have been stored in accordance with the following:

  * Prospective Fresh:

    * Room temperature (15 °C to 25 °C) for ≤24 hrs
    * Refrigerated (2 °C to 8 °C) for ≤ 7 days
  * Prospective Frozen:

    * -15 ºC to -25 ºC for ≤ 2 months
    * -60 ºC to -90 ºC for ≤ 4 months
  * Retrospective Archived:

    * Frozen
* At the time of QIAstat-Dx testing, specimen must not have undergone more than three (3) freeze/thaw cycles.
* Prospective Samples Only: Specimen must have been collected on or after the date of prospective study activation at the Clinical collection and testing site.
* Retrospective Samples Only: Specimens must have a positive diagnosis as per Standard of Care for any of the following viral targets:

Herpes simplex virus 1 (HSV-1) Herpes simplex virus 2 (HSV-2) Human herpesvirus 6 (HHV-6) Human parechovirus (HPeV) Varicella zoster virus (VZV) Cytomegalovirus (CMV)

Exclusion Criteria:

* Residual CSF specimen has been centrifuged.
* Residual CSF specimen subject identification or label is unclear or missing.
* Residual CSF specimen container has obvious physical damage.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with signs and symptoms of Meningitis/Encephalitis infection
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
PPA | 7 months
  Positive percent agreement
NPA | 7 months
  Negative percent agreement

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, Principal Investigator — Qiagen Manchester Limited
Locations (1):
- QIAGEN, Manchester, United Kingdom